CLINICAL TRIAL: NCT05823064
Title: Respiratory Morbidities and Outcome in Late Preterm in Neonatal ICU of Assiut University Children Hospital, One Year Study
Brief Title: Respiratory Morbidities and Outcome in Late Preterm in Neonatal ICU
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Nady Sadik, principal investigator, Assiut University
Other Study IDs: Respiratory morbidities
Record Dates: First submitted 2023-04-10; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Respiratory Morbidities

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
Aim of the work:

To assess the respiratory morbidities & outcomes in late preterm infants in the neonatal ICU of Assiut university children's Hospital.

DETAILED DESCRIPTION:
In the world, Preterm birth rates continue to rise. Many reasons account for this increase, such as demographic changes, infertility treatments, increases in maternal age, more multiple gestations, increasing obesity rates, and maternal comorbid conditions.

To evaluate the occurrence and impact of a condition, a precise definition and its related outcomes are necessary. Thus, a general classification for selected gestational age categories has been reported. Preterm birth refers to all deliveries < 37-0/7 weeks; this classification includes very preterm (< 32-0/7 weeks), moderately preterm (32-0/7 to 33-6/7 weeks), and late preterm births (34-0/7 to 36-6/7 weeks). Term births refer to deliveries that occur from 37-0/7 to 42-0/7 weeks, and post-term births refer to any delivery occurring after 42-0/7 weeks.

Neonates born between 34 and 36 weeks of gestation (late preterm or near-term births) comprise 71% of all preterm births in the United States.

Late preterm neonates have significantly higher rates of morbidity and mortality relative to those born at term (37-42 weeks).

In addition to higher risks for serious health complications, the mortality rate for late preterm infants is 3-fold higher than that for term infants (7.7 vs 2.5 per 1000 live births).

Late preterm delivery (71% of all preterm births) increases the incidence of respiratory pathology as respiratory distress syndrome (RDS), Transient tachypnea of the newborn (TTN), pneumonia with chest x-ray verification, persistent apnea and bradycardia, pulmonary hypertension, pneumothorax, meconium aspiration, pulmonary hypoplasia,( respiratory failure ) and the need of ventilator support when compared to term delivery.

Late preterm newborns increase other risks for feeding difficulty, jaundice, hypoglycemia, temperature instability, apnea, and respiratory distress.

ELIGIBILITY:
Inclusion Criteria:

* late preterm neonates admitted to the Neonatal intensive care unit (NICU) at Assiut University Children's Hospital for one year.

Exclusion Criteria:

patients with congenital heart diseases and multiple congenital anomalies.

Ages: 1 Day to 28 Days | Sex: All
Age Groups: Child
Study Population: 20 Neonates born between 34 and 36 weeks of gestation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
To assess the respiratory morbidities | base line
  To assess the respiratory morbidities in late preterm infants in neonatal ICU of Assiut university children hospital .

CONTACTS AND LOCATIONS:
Overall Officials: Nafisa H Refaat, Principal Investigator — Assiut University; Mohamed A Sayed, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided